CLINICAL TRIAL: NCT01261611
Title: A Phase III, Randomised, Double-blind and Open Label Phase, Active and Placebo Controlled Study Comparing the Short-term Efficacy of Two Formulations of Clostridium Botulinum Type A Toxin (Dysport and Dysport NG) to Placebo, and Assessing the Short and Long Term Efficacy and Safety of Dysport NG Following Repeated Treatments of Subjects With Cervical Dystonia
Brief Title: Study Comparing Short Term Efficacy of Dysport and Dysport NG to Placebo, and to Assess Efficacy and Safety of Dysport NG of Subjects With Cervical Dystonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Y-52-52120-134; 2010-019907-43 (EudraCT Number)
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dysport NG (Experimental): 500U (1mL) administered as intramuscular injection on day 1 of treatment cycle 1 and 2.
  250U (0.5mL), 500U (1mL) or 750U (1.5mL) administered as intramuscular injection on day 1 of treatment cycle 3.
  250U (0.5mL), 500U (1mL), 750U (1.5mL) or 1000U (2mL) administered as intramuscular injection on day 1 of treatment cycle 4 and 5.
  Interventions: Biological: Botulinum toxin type A
- Dysport (Active Comparator): 500U (1mL) injected as intramuscular injection on day 1 of treatment cycle 1.
  Interventions: Biological: Botulinum toxin type A
- Placebo (Placebo Comparator): 1mL administered as, intramuscular injection on day 1 of treatment cycle 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — I.M. (in the muscle) injection on day 1 of up to 5 treatment cycles.
  Other Names: AbobotulinumtoxinA (DysportRU®)
  Arms: Dysport NG
Biological: Botulinum toxin type A — I.M. injection on day 1 of treatment cycle 1.
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: Dysport
Drug: Placebo — I.M. injection on day 1 of treatment cycle 1.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate how well a new drug called Dysport NG works and how safe it is, when it is used for the treatment of cervical dystonia. Dysport NG will be compared to an approved drug called Dysport.

DETAILED DESCRIPTION:
The primary study objectives will be assessed in terms of improvement of the subject's CD at a pre-defined time point after treatment. The primary study objectives are to demonstrate the superiority of Dysport NG to placebo in terms of efficacy and to test the non-inferior efficacy of Dysport NG, when compared to Dysport, in CD subjects. In addition to testing for the primary study objectives, the superiority in terms of efficacy of Dysport versus placebo, will be assessed.

This clinical study was designed and implemented and reported in accordance with the International Conference on Harmonization (ICH) Harmonized Tripartite Guidelines for Good Clinical Practice (GCP), with applicable local regulations (including European Directive 2001/20/EC, US Code of Federal Regulations Title 21, and with the ethical principles laid down in the Declaration of Helsinki.

A large body of evidence demonstrates the safety and efficacy of Dysport across several clinical indications. This study was the first use of Dysport NG in humans with CD. The active substance (BTX-A-HAC) in Dysport NG was the same as in the currently marketed Dysport product and had the same mechanism of action. Dysport NG was, therefore, expected to have the same efficacy and safety profile in humans as Dysport, with the advantage of eliminating the potential risk of transmission of infective agents, by the substitution of plant and synthetic products for human and animal-derived products. However, due to the change of excipient, thorough assessment of the safety and efficacy of Dysport NG is necessary. Previous clinical studies indicate that the maximum effect of Dysport and maximum improvements in CD are observed approximately 4 weeks post treatment, after which there is a gradual return to baseline disease status. The Week 4 follow up visit after the first treatment cycle was therefore, chosen as the primary time point of interest. Retreatment is necessary in order to maintain the beneficial effect and the long term treatment of CD. Previously conducted long term studies demonstrate the maintenance of the therapeutic effect of Dysport following repeated treatments, with a favourable short and long term safety and immunogenicity profile.

ELIGIBILITY:
Inclusion Criteria:

* Dystonia with at least 18 months duration since onset.
* Previously untreated with Botulinum toxin-A (BTX-A) or -B or a minimum of 14 weeks since the last injection.
* TWSTRS score at baseline of: Total score ≥ 30, Severity Sub-Scale score ≥ 15, Disability Sub-Scale score ≥ 3, Pain Sub-Scale score ≥ 2.

Exclusion Criteria:

* Known hypersensitivity to Botulinum toxin (BTX) or related compounds or any component in the study drug formulation (including cow milk protein).
* Pure anterocollis or pure retrocollis.
* In apparent remission from Cervical Dystonia.
* Known clinically significant underlying swallowing or respiratory abnormality which might be exacerbated by BTX treatment.
* Previous poor response to BTX treatment or known presence of BTX neutralising antibodies.
* Previous phenol or alcohol injections into the neck muscles.
* Previous myotomy or denervation surgery involving the neck or shoulder region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (57):
- Australia (4):
  - Monash Medical Centre, Clayton
  - Austin Hospital, Heidelberg
  - Department of Neurosciences Alfred Hospital, Prahran
  - Westmead Hospital, Westmead
- Austria (2):
  - Univ.-Klinik für Neurologie, Innsbruck
  - Univ.-Klinik für Neurologie, Vienna
- Belgium (5):
  - AZ St. Jan, Bruges
  - Universitair Ziekenhuis Antwerpen, Edegem
  - AZ Sint Lucas, Ghent
  - Centre Hospitalier Universitaire de Liège, Liège
  - HH Ziekenhuis, Roeselare
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Pardubicka krajska nemocnice, Pardubice
  - RESEARCH SITE s.r.o., Pilsen
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (6):
  - CHU Amiens, Amiens
  - Hopital Neurologique, Bron
  - CHU Caremeau, Nîmes
  - CHU Bordeaux, Pessac
  - CHU Strasbourg, Strasbourg
  - Hopital Purpan, Toulouse
- Germany (10):
  - Neurologische Klinik u. Poliklinik, Berlin
  - Neurologische Klinik u. Poliklinik, Bonn
  - Neurologische Klinik, Düsseldorf
  - Neurologische Klinik, Halle
  - Neurologische Klinik, Hanover
  - Neurologische Klinik, Leipzig
  - Neurologische Klinik, München
  - Neurologische Klinik, Tübingen
  - Neurologische Klinik, Wiesbaden
  - Neurologische Klinik, Würzburg
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Jósa András Oktató Kórház Nonprofit Kft., Nyíregyháza
  - Pécsi Tudományegyetem, Pécs
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
- Poland (6):
  - Pomorskie Centrum Traumatologii im. M. Kopernika w Gdansku, Gdansk
  - Specjalistyczna Praktyka Lekarska, Katowice
  - Malopolskie Centrum Medyczne, Krakow
  - Gabinet Lekarski, Lodz
  - Niepubliczny Zaklad Opieki Zdrowotnej, Poznan
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
- Portugal (2):
  - Hospital Santa Maria, Lisbon
  - Hospital Geral de Santo Antonio, Porto
- Russia (6):
  - Research Medical Complex "Vashe Zdorovie", Kazan'
  - Research Center of Neurology of RAMS, Moscow
  - Nizhniy Novgorod Research Institute for Traumatology and Orthopaedics, Nizhny Novgorod
  - Russian Medical Military Academy n.a. S.M.Kirov, Saint Petersburg
  - Samara Regional Clinical Hospital, Samara
  - Smolensk State Medical Academy Smolensk Regional Clinical Hospital, Smolensk
- Ukraine (8):
  - Bukovinian Medical State University, Chernivtsi
  - Ukrainian State Institute of Medical and Social Problems of Disability, Dnipropetrovsk
  - Donetsk Railroad Clinical Hospital, Donetsk
  - Institute of Neurology, Psychiatry and Narcology AMS of Ukraine, Kharkiv
  - Lviv Regional Clinical Hospital, Lviv
  - Municipal Institution "Odesa Regional Clinical Hospital", Odesa
  - Uzhgorod National University, Uzhhorod
  - Vinnytsya National Medical University, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Poewe W, Burbaud P, Castelnovo G, Jost WH, Ceballos-Baumann AO, Banach M, Potulska-Chromik A, Ferreira JJ, Bihari K, Ehler E, Bares M, Dzyak LA, Belova AN, Pham E, Liu WJ, Picaut P. Efficacy and safety of abobotulinumtoxinA liquid formulation in cervical dystonia: A randomized-controlled trial. Mov Disord. 2016 Nov;31(11):1649-1657. doi: 10.1002/mds.26760. Epub 2016 Sep 21. PMID 27653448

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited at 61 centres in Australia (2 subjects), Austria (9 subjects), Belgium (9 subjects), Czech Republic (58 subjects), France (31 subjects), Germany (38 subjects), Hungary (44 subjects), Poland (68 subjects), Portugal (12 subjects), Russia (36 subjects) and Ukraine (62 subjects).
Pre-assignment Details: 382 subjects screened, 369 randomised due to 13 screen failures.
Groups:
- Dysport NG: Up to 5 treatment cycles of Dysport NG
- Dysport: 1 treatment cycle of Dysport
- Placebo: 1 treatment cycle of placebo
Period: Treatment Cycle 1
Arm/Group | Dysport NG | Dysport | Placebo
Started | 156 | 159 | 54
Completed | 152 | 156 | 52
Not Completed | 4 | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 2
Period: Treatment Cycle 2
Arm/Group | Dysport NG | Dysport | Placebo
Started | 359 (All but 1 who completed DB period entered the open label period. This subject remained at Cycle 1.) | 0 | 0
Completed | 346 | 0 | 0
Not Completed | 13 | 0 | 0
Not completed — Completed study | 4 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Not otherwise specified | 2 | 0 | 0
Period: Treatment Cycle 3
Arm/Group | Dysport NG | Dysport | Placebo
Started | 346 | 0 | 0
Completed | 316 | 0 | 0
Not Completed | 30 | 0 | 0
Not completed — Completed study | 24 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Treatment Cycle 4
Arm/Group | Dysport NG | Dysport | Placebo
Started | 316 | 0 | 0
Completed | 220 | 0 | 0
Not Completed | 96 | 0 | 0
Not completed — Completed study | 87 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Not otherwise specified | 3 | 0 | 0
Period: Treatment Cycle 5
Arm/Group | Dysport NG | Dysport | Placebo
Started | 220 | 0 | 0
Completed | 217 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dysport NG: 500U (1mL) administered as intramuscular injection on day 1 of treatment cycle 1 and 2.
  250U (0.5mL), 500U (1mL) or 750U (1.5mL) administered as intramuscular injection on day 1 of treatment cycle 3.
  250U (0.5mL), 500U (1mL), 750U (1.5mL) or 1000U (2mL) administered as intramuscular injection on day 1 of treatment cycle 4 and 5.
  Botulinum type A toxin (Dysport NG): I.M. (in the muscle) injection on day 1 of up to 5 treatment cycles.
- Dysport: 500U (1mL) injected as intramuscular injection on day 1 of treatment cycle 1.
  Botulinum type A toxin (Dysport®): I.M. injection on day 1 of treatment cycle 1.
- Total: Total of all reporting groups
Arm/Group | Dysport NG | Dysport | Placebo | Total
Number analyzed (Participants) | 156 | 159 | 54 | 369
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (12.4) | 49.1 (12.0) | 49.7 (10.8) | 50.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 101 | 34 | 235
  Male | 56 | 58 | 20 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 154 | 154 | 49 | 357
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 3 | 9
Time since diagnosis of CD, years [Mean (Standard Deviation); unit: years] | 7.13 (7.95) | 6.88 (7.49) | 6.25 (7.31) | 6.84 (7.63)
Baseline Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Total score [Mean (Standard Deviation); unit: Units on a scale] — TWSTRS measures the degree of CD and is comprised of three different components, namely Severity, Disability and Pain subscales. There is an ordinal scale score and range for each component. Severity scores range from 0 (absence of severity) to 35 (maximum severity), Disability scores range from 0 (no disability) to 30 (maximum disability) and Pain scores range from 0 (no pain) to 20 (maximum pain). TWSTRS Total score is the sum of the 3 component scores ranging from 0 to a maximum of 85, with higher scores denoting worse outcome.
  Units on a scale | 44.56 (9.20) | 46.23 (8.82) | 47.02 (9.19) | 45.64 (9.06)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Total Score Following First Treatment Cycle
Description: TWSTRS measures the degree of CD and is comprised of three different components, namely Severity, Disability and Pain subscales. There is an ordinal scale score and range for each component. Severity scores range from 0 (absence of severity) to 35 (maximum severity), Disability scores range from 0 (no disability) to 30 (maximum disability) and Pain scores range from 0 (no pain) to 20 (maximum pain). TWSTRS Total score is the sum of the 3 component scores ranging from 0 to a maximum of 85, with higher scores denoting worse outcome. If the change from baseline is negative, this represents an improvement in symptoms.
Time Frame: Baseline and Week 4
Population: Analysis based on number (n) of subjects in the Intent to Treat (ITT) population (all randomised subjects who received at least one injection of study treatment regardless of the amount of study treatment administered). The ITT population was analysed using subjects as randomised. Missing data were not imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Dysport NG; Dysport: 500U
Arm/Group | Dysport NG | Dysport | Placebo
Number analyzed (Participants) | 153 | 156 | 53
Units on a scale | -12.46 [-14.30 to -10.62] | -13.99 [-15.78 to -12.21] | -3.93 [-6.74 to -1.12]
Statistical Analysis 1: Comparison: Dysport NG vs Placebo; A pre-specified analysis of the LS mean difference between the Dysport NG and Placebo arms was performed. A total of 210 subjects were included in the analysis; Test type: Superiority or Other; p < 0.0001, ANCOVA; An ANCOVA on the change from baseline, baseline TWSTRS Total score, baseline BTX status and pooled centre as explanatory variables was performed
Statistical Analysis 2: Comparison: Dysport vs Placebo; A pre-specified analysis of the LS mean difference between the Dysport and Placebo arms was performed. A total of 213 subjects were included in the analysis; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dysport NG vs Dysport; A pre-specified analysis of the LS mean difference between the Dysport NG and Dysport arms was performed. A total of 315 subjects were included in the analysis; Test type: Non-Inferiority or Equivalence — An ANCOVA on the change from baseline with treatment, baseline TWSTRS Total score, BTX status at baseline and pooled centre as explanatory variables had been performed. The non-inferiority margin was 3 points; LS mean difference = 1.532, 95% CI 2-sided [-0.819 to 3.883]

2. Secondary Outcome: Change From Baseline in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Severity Subscale Score Following First Treatment Cycle
Description: TWSTRS measures the degree of CD and comprises three different components, one of which is the Severity subscale. TWSTRS Severity subscale scores range from 0 (absence of severity) to 35 (maximum severity). If the change from baseline is negative, this represents an improvement in symptoms.
Time Frame: Baseline and Week 4
Population: Analysis based on number (n) of subjects in the ITT population (all randomised subjects who received at least one injection of study treatment regardless of the amount of study treatment administered). The ITT population was analysed using subjects as randomised. Missing data were not imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Dysport NG | Dysport | Placebo
Number analyzed (Participants) | 153 | 156 | 53
Units on a scale | -6.2 [-7.0 to -5.4] | -6.6 [-7.3 to -5.8] | -1.9 [-3.1 to -0.6]

3. Secondary Outcome: Change From Baseline in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Disability Subscale Score Following First Treatment Cycle
Description: TWSTRS measures the degree of CD and comprises three different components, one of which is the Disability subscale. TWSTRS Disability subscale scores range from 0 (no disability) to 30 (maximum disability). If the change from baseline is negative, this represents an improvement in symptoms.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Dysport NG | Dysport | Placebo
Number analyzed (Participants) | 153 | 156 | 53
Units on a scale | -3.3 [-4.1 to -2.6] | -3.9 [-4.7 to -3.2] | -0.8 [-1.9 to 0.4]

4. Secondary Outcome: Change From Baseline in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Pain Subscale Score Following First Treatment Cycle
Description: TWSTRS measures the degree of CD and comprises three different components, one of which is the Pain subscale. TWSTRS Pain subscale scores range from 0 (no pain) to 20 (maximum pain). If the change from baseline is negative, this represents an improvement in symptoms.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Dysport NG | Dysport | Placebo
Number analyzed (Participants) | 153 | 156 | 53
Units on a scale | -3.10 [-3.70 to -2.51] | -3.44 [-4.03 to -2.86] | -1.21 [-2.12 to -0.29]

5. Secondary Outcome: Change From Baseline in Subject Visual Analogue Score (VAS) for Pain From Cervical Dystonia Following First Treatment Cycle
Description: The assessment was made on a continuous 100-mm horizontal line with a scale range of 0 mm (no pain) to 100 mm (worst possible pain).
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Dysport NG | Dysport | Placebo
Number analyzed (Participants) | 153 | 156 | 53
Units on a scale | -14.8 [-19.0 to -10.7] | -19.2 [-23.3 to -15.2] | -3.4 [-9.8 to 3.0]

6. Secondary Outcome: Change From Baseline in Subject Visual Analogue Score (VAS) for Symptoms of Cervical Dystonia Following First Treatment Cycle
Description: The assessment was made on a continuous 100-mm horizontal line with a scale range of 0 mm (no symptoms) to 100 mm (worst possible symptoms).
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Dysport NG | Dysport | Placebo
Number analyzed (Participants) | 152 | 156 | 53
Units on a scale | -18.7 [-22.7 to -14.7] | -23.6 [-27.5 to -19.7] | -3.3 [-9.4 to 2.8]

7. Secondary Outcome: Percentage of Treatment Responders Following First Treatment Cycle
Description: A treatment responder was defined as a patient with >30% improvement in TWSTRS Total score compared to baseline.
  TWSTRS measures the degree of CD and is comprised of three different components, namely Severity, Disability and Pain subscales. There is an ordinal scale score and range for each component. Severity scores range from 0 (absence of severity) to 35 (maximum severity), Disability scores range from 0 (no disability) to 30 (maximum disability) and Pain scores range from 0 (no pain) to 20 (maximum pain). TWSTRS Total score is the sum of the 3 component scores ranging from 0 to a maximum of 85, with higher scores denoting worse outcome. If the change from baseline is negative, this represents an improvement in symptoms.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Dysport NG | Dysport | Placebo
Number analyzed (Participants) | 153 | 156 | 53
Percentage of participants | 45.8 | 55.8 | 20.8

8. Secondary Outcome: Change From Baseline in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Total Score for Treatment Cycles 2 to 5
Description: as for outcome 1
Time Frame: Treatment cycle Baseline and Week 4
Population: Analysis based on number (n) of subjects in the ITT population (all randomised subjects who received at least one injection of study treatment regardless of the amount of study treatment administered) in each cycle. The ITT population was analysed using subjects as randomised. Missing data were not imputed.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Dysport NG: All doses
Arm/Group | Dysport NG
Number analyzed (Participants) | 359
Units on a scale
  Cycle 2: number analyzed (Participants) | 349
  Cycle 2 | -15.35 [-16.36 to -14.34]
  Cycle 3: number analyzed (Participants) | 345
  Cycle 3 | -14.85 [-15.86 to -13.84]
  Cycle 4: number analyzed (Participants) | 312
  Cycle 4 | -15.58 [-16.61 to -14.55]
  Cycle 5: number analyzed (Participants) | 219
  Cycle 5 | -15.28 [-16.42 to -14.14]

9. Secondary Outcome: Change From Baseline in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Severity Score for Treatment Cycles 2 to 5
Description: as for outcome 2
Time Frame: Treatment cycle Baseline and Week 4
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Dysport NG
Number analyzed (Participants) | 359
Units on a scale
  Cycle 2: number analyzed (Participants) | 349
  Cycle 2 | -7.2 [-7.6 to -6.7]
  Cycle 3: number analyzed (Participants) | 345
  Cycle 3 | -7.1 [-7.5 to -6.6]
  Cycle 4: number analyzed (Participants) | 312
  Cycle 4 | -7.3 [-7.7 to -6.8]
  Cycle 5: number analyzed (Participants) | 219
  Cycle 5 | -7.0 [-7.5 to -6.4]

10. Secondary Outcome: Change From Baseline in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Disability Score for Treatment Cycles 2 to 5
Description: as for outcome 3
Time Frame: Treatment cycle Baseline and Week 4
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Dysport NG
Number analyzed (Participants) | 359
Units on a scale
  Cycle 2: number analyzed (Participants) | 349
  Cycle 2 | -4.7 [-5.2 to -4.3]
  Cycle 3: number analyzed (Participants) | 345
  Cycle 3 | -4.6 [-5.0 to -4.1]
  Cycle 4: number analyzed (Participants) | 312
  Cycle 4 | -5.0 [-5.5 to -4.5]
  Cycle 5: number analyzed (Participants) | 219
  Cycle 5 | -4.9 [-5.5 to -4.3]

11. Secondary Outcome: Change From Baseline in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Pain Subscale Score for Treatment Cycles 2 to 5
Description: as for outcome 4
Time Frame: Treatment cycle Baseline and Week 4
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Dysport NG
Number analyzed (Participants) | 359
Units on a scale
  Cycle 2: number analyzed (Participants) | 349
  Cycle 2 | -3.45 [-3.8 to -3.1]
  Cycle 3: number analyzed (Participants) | 345
  Cycle 3 | -3.21 [-3.57 to -2.85]
  Cycle 4: number analyzed (Participants) | 312
  Cycle 4 | -3.34 [-3.69 to -2.98]
  Cycle 5: number analyzed (Participants) | 219
  Cycle 5 | -3.41 [-3.79 to -3.04]

12. Secondary Outcome: Change From Baseline in Subject Visual Analogue Score (VAS) for Pain From Cervical Dystonia for Treatment Cycles 2 to 5
Description: as for outcome 5
Time Frame: Treatment cycle Baseline and Week 4
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Dysport NG
Number analyzed (Participants) | 359
Units on a scale
  Cycle 2: number analyzed (Participants) | 349
  Cycle 2 | -20.1 [-22.5 to -17.6]
  Cycle 3: number analyzed (Participants) | 345
  Cycle 3 | -17.8 [-20.4 to -15.2]
  Cycle 4: number analyzed (Participants) | 311
  Cycle 4 | -18.0 [-20.5 to -15.4]
  Cycle 5: number analyzed (Participants) | 219
  Cycle 5 | -16.1 [-19.3 to -12.8]

13. Secondary Outcome: Change From Baseline in Subject Visual Analogue Score (VAS) for Symptoms of Cervical Dystonia for Treatment Cycles 2 to 5
Description: The assessment was made on a continuous 100-mm horizontal line with a scale of 0 mm (no symptoms) to 100 mm (worst possible symptoms).
Time Frame: Treatment cycle Baseline and Week 4
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Dysport NG
Number analyzed (Participants) | 359
Units on a scale
  Cycle 2: number analyzed (Participants) | 349
  Cycle 2 | -24.0 [-26.4 to -21.7]
  Cycle 3: number analyzed (Participants) | 345
  Cycle 3 | -18.9 [-21.4 to -16.4]
  Cycle 4: number analyzed (Participants) | 311
  Cycle 4 | -21.0 [-23.5 to -18.5]
  Cycle 5: number analyzed (Participants) | 219
  Cycle 5 | -18.2 [-21.2 to -15.2]

14. Secondary Outcome: Percentage of Treatment Responders for Treatment Cycles 2 to 5
Description: as for outcome 7
Time Frame: Treatment cycle Baseline and Week 4
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Dysport NG
Number analyzed (Participants) | 359
Percentage of participants
  Cycle 2: number analyzed (Participants) | 349
  Cycle 2 | 58.5
  Cycle 3: number analyzed (Participants) | 345
  Cycle 3 | 56.8
  Cycle 4: number analyzed (Participants) | 312
  Cycle 4 | 63.5
  Cycle 5: number analyzed (Participants) | 219
  Cycle 5 | 57.5

ADVERSE EVENTS:
Time Frame: 2 years
Description: Analysis based on number of subjects in the safety population (all randomised subjects who received at least one injection of study treatment). One subject was randomised to Dysport 500 U but actually received placebo; therefore, this subject was counted in the placebo group for the safety population analysis (n=55 not n=54). Data are broken down by dose across all treatment cycles and the denominator (total number of patients at risk) for each group could not be reported in participant flow.
Groups:
- Dysport NG, 250U; Dysport NG, 500U; Dysport NG, 750U; Dysport NG, 1000U: Subjects in the safety population were analysed as treated.
- Dysport, 500U; Placebo: The safety population was analysed using subjects as treated. One subject was randomised to Dysport 500 U but actually received placebo; therefore, this subject was counted in the placebo group for the safety population, and the Dysport group for the ITT population.
Arm/Group | Dysport NG, 250U | Dysport NG, 500U | Dysport NG, 750U | Dysport NG, 1000U | Dysport, 500U | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 16/363 | 3/210 | 1/57 | 3/156 | 0/55
Other Adverse Events (participants affected / at risk) | 1/4 | 59/363 | 29/210 | 7/57 | 15/156 | 1/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dysport NG, 250U (N=4) | Dysport NG, 500U (N=363) | Dysport NG, 750U (N=210) | Dysport NG, 1000U (N=57) | Dysport, 500U (N=156) | Placebo (N=55)
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Paget-Schroetter syndrome (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Proctitis infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thyroid cyst (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesphageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport NG, 250U (N=4) | Dysport NG, 500U (N=363) | Dysport NG, 750U (N=210) | Dysport NG, 1000U (N=57) | Dysport, 500U (N=156) | Placebo (N=55)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 38 (54) | 20 (25) | 5 (5) | 11 (11) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 21 (26) | 9 (9) | 2 (2) | 4 (4) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 11 (15) | 13 (14) | 6 (6) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No